CLINICAL TRIAL: NCT04356196
Title: Comparative Study Between the Efficacy of Verapamil and Bisoprolol on Reduction of Bleeding During Endoscopic Sinus Surgery Under General Anaesthesia.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Ali Hassan Refaat AL-Quossi, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Verapamil, Bisoprolol in ESS
Record Dates: First submitted 2020-04-18; First posted 2020-04-22 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Endoscopic Sinus Surgery; Heart Rate; Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Verapamil; Bisoprolol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verapamil group (Experimental): 45 patients will receive 80 mg oral verapamil 3 hours pre-operative
  Interventions: Drug: Verapamil
- Bisoprolol group (Experimental): 45 patients will receive Bisoprolol 5mg PO 3 hours preoperative
  Interventions: Drug: Bisoprolol
- placebo group (Experimental): 45 patients will receive placebo tablet PO 3 hours preoperative .
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Verapamil — Verapamil is a phenylalkylamine calcium channel blocker used in the treatment of high blood pressure, heart arrhythmias, and angina
  Other Names: Isoptin
  Arms: Verapamil group
Drug: Bisoprolol — Bisoprolol is a cardioselective β1-adrenergic blocking agent used to treat high blood pressure.
  Other Names: concor
  Arms: Bisoprolol group
Drug: Placebo oral tablet — Placebo oral tablet
  Arms: placebo group

SUMMARY:
The study aims to compare the effect of addition of verapamil and Bisoprolol to general anasthesia aimed reduction in heart rate and blood loss during endoscopic sinus surgery.

DETAILED DESCRIPTION:
Intra-operative bleeding presents a larger obstacle to endoscopic visualization. Blood obscures the anatomy of the surgical field and dirties the endoscope lens causing greater difficulty with visualization. This situation increases the risk of complications, including brain injury, orbital or optic nerve injury, and catastrophic bleeding from major vessels (e.g., internal carotid artery) 1.

Endoscopic sinus surgery (ESS) is a minimally invasive technique used to restore sinus ventilation and function in patients with recurrent acute or chronic infective sinusitis in whom medical therapy has failed. The term ESS is used to draw attention to the potential for reestablishing natural mucociliary clearance mechanism, drainage and aeration of sinuses, whilst maintaining as much of the normal anatomy as possible. Over last few years this technique has become popular worldwide due to its minimally invasive nature and preservation of mucosa2.

Continued bleeding into the surgical field during ESS not only impairs endoscopic vision but can lead to complications3. Compared with conventional anesthesia, total intravenous anesthesia (TIVA) has been previously reported to result in reduced blood loss when used for FESS. However, few recent studies point out that TIVA may not significantly reduce blood loss 4-5.

Controlled hypotension has been used to reduce bleeding and the need for blood transfusions, and provide a satisfactory bloodless surgical field . Controlled hypotension is defined as a reduction of the systolic blood pressure to 80-90 mm Hg, a reduction of mean arterial pressure (MAP) to 50-65 mm Hg or a 30% reduction of baseline MAP 6. The physiological principle which underlies hypotensive anesthesia is a natural survival mechanism. When profuse bleeding occurs, the blood pressure drops. This drop leads to a reduction or cessation of the bleeding, blood pressure stabilization, and recovery. Accordingly, reducing the patient's blood pressure during surgery can potentially reduce

overall bleeding. Since bleeding in the surgical field is also reduced, the surgical field operating conditions are improved 7 .

Pharmacological agents used for controlled hypotension include those agents that can be used successfully alone and those that are used adjunctively to limit dosage requirements and, therefore, the adverse effects of the other agents. Agents used successfully alone include inhalation anaesthetics, sodium nitroprusside, nitroglycerin, trimethaphan camsilate, alprostadil (prostaglandin E1), adenosine, remifentanil, and agents used in spinal anaesthesia. Agents that can be used alone or in combination include calcium channel antagonists (e.g. nicardipine), beta-adrenoceptor antagonists (beta- blockers) [e.g. bisoprolo, propranolol, esmolol] and fenoldopam. Agents that are mainly used adjunctively include ACE inhibitors and clonidine. New agents and techniques have been recently evaluated for their ability to induce effective hypotension without impairing the perfusion of vital organs 8.

Calcium channel blockers are drugs that block the entry of calcium into the muscle cells of the heart and arteries. Thus, by blocking the entry of calcium, calcium channel blockers reduce electrical conduction within the heart, decrease the force of contraction (work) of the muscle cells, and dilate arteries which reduces blood pressure and thereby the effort the heart must exert to pump blood 9.

Although calcium channel blockers have a similar mechanism of action, they differ in their ability to affect heart muscle vs. arteries, and they differ in their ability to affect heart rate and contraction. For example; verapamil (Covera-HS, Verelan PM, Calan), reduces the strength and rate of the heart's contraction and are used in treating abnormal heart rhythms10.

Beta-blockers antagonise the effects of sympathetic nerve stimulation or circulating catecholamines at beta-adrenoceptors which are widely distributed throughout body systems. Beta1-receptors are predominant in the heart (and kidney) while beta2- receptors are predominant in other organs such as the lung, peripheral blood vessels and skeletal muscle11.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years.
* patients of both genders.
* ASA grade I - II.

Exclusion Criteria:

* Patient refusal.
* Any contraindication of B- blocker:

  1. Athma , COPD
  2. Bradycardia , Heart block
  3. Acute decompensated heart failure
  4. Peripheral vascular disease
* Any contraindication of calcium channel blocker:

  1. AV conduction defects (2nd and 3rd degree AV block).
  2. Sick sinus syndrome .
  3. Wolf-Parkinson-White Syndrome.
  4. History of congestive heart failure.
  5. Patients on long-term ß-blocker therapy.
  6. Patients with allergy to medication included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | intraoperative
  heart beats for minutes
Estimated Blood Loss | end of operation assessment
  Estimated blood loss in milliliters per hour is calculated by subtracting the volume of total irrigation used during the case from the total amount of fluid in the suction canister at the end of surgery dividing by surgical time in hours.

SECONDARY OUTCOMES:
The Boezaart and van der Merwe intraoperative surgical field scale | Every 15 minutes for the duration of surgery
  Boezaart Bleeding Scale (BBS) (0 - no bleeding (cadaveric conditions), 1 - Slight bleeding, no suctioning required, 2 - Slight bleeding, occasional suctioning required, 3 - Slight bleeding, frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed, 4 - Moderate bleeding, frequent suctioning required, and bleeding threatens surgical field directly after suction is removed, 5 - Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible).
plasma norepinephrine concentrations | baseline before Anastasia ( in the holding area with insertion of I.V. cannula) and three hours after the end of surgery.
  plasma norepinephrine concentrations measured by enzyme immunoassay as venous blood samples about 4ml will be collected from each patient under aseptic condition
serum cortisol concentrations | baseline before Anastasia ( in the holding area with insertion of I.V. cannula) and three hours after the end of surgery.
  serum cortisol will be measured by enzyme immunoassay as venous blood samples about 4ml will be collected from each patient under aseptic condition

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Sayed Hassanein, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Thongrong C, Kasemsiri P, Carrau RL, Bergese SD. Control of bleeding in endoscopic skull base surgery: current concepts to improve hemostasis. ISRN Surg. 2013 Jun 13;2013:191543. doi: 10.1155/2013/191543. Print 2013. PMID 23844295
- [Background] Hadad G, Bassagasteguy L, Carrau RL, Mataza JC, Kassam A, Snyderman CH, Mintz A. A novel reconstructive technique after endoscopic expanded endonasal approaches: vascular pedicle nasoseptal flap. Laryngoscope. 2006 Oct;116(10):1882-6. doi: 10.1097/01.mlg.0000234933.37779.e4. PMID 17003708
- [Background] Stammberger H. Endoscopic endonasal surgery--concepts in treatment of recurring rhinosinusitis. Part II. Surgical technique. Otolaryngol Head Neck Surg. 1986 Feb;94(2):147-56. doi: 10.1177/019459988609400203. PMID 3083327
- [Background] Stankiewicz JA, Lal D, Connor M, Welch K. Complications in endoscopic sinus surgery for chronic rhinosinusitis: a 25-year experience. Laryngoscope. 2011 Dec;121(12):2684-701. doi: 10.1002/lary.21446. Epub 2011 Nov 15. PMID 22086769
- [Background] Eberhart LH, Folz BJ, Wulf H, Geldner G. Intravenous anesthesia provides optimal surgical conditions during microscopic and endoscopic sinus surgery. Laryngoscope. 2003 Aug;113(8):1369-73. doi: 10.1097/00005537-200308000-00019. PMID 12897561
- [Background] Ankichetty SP, Ponniah M, Cherian V, Thomas S, Kumar K, Jeslin L, Jeyasheela K, Malhotra N. Comparison of total intravenous anesthesia using propofol and inhalational anesthesia using isoflurane for controlled hypotension in functional endoscopic sinus surgery. J Anaesthesiol Clin Pharmacol. 2011 Jul;27(3):328-32. doi: 10.4103/0970-9185.83675. PMID 21897501
- [Background] Degoute CS, Ray MJ, Manchon M, Dubreuil C, Banssillon V. Remifentanil and controlled hypotension; comparison with nitroprusside or esmolol during tympanoplasty. Can J Anaesth. 2001 Jan;48(1):20-7. doi: 10.1007/BF03019809. PMID 11212044
- [Background] Tobias JD. Controlled hypotension in children: a critical review of available agents. Paediatr Drugs. 2002;4(7):439-53. doi: 10.2165/00128072-200204070-00003. PMID 12083972
- [Background] Degoute CS. Controlled hypotension: a guide to drug choice. Drugs. 2007;67(7):1053-76. doi: 10.2165/00003495-200767070-00007. PMID 17488147